CLINICAL TRIAL: NCT02932618
Title: A Phase 3, Prospective, Multicenter, Uncontrolled, Open-Label Clinical Study to Determine the Efficacy, Safety, and Tolerability of rVWF With or Without ADVATE in the Treatment and Control of Bleeding Episodes, the Efficacy and Safety of rVWF in Elective and Emergency Surgeries, and the Pharmacokinetics (PK) of rVWF in Children Diagnosed With Severe Von Willebrand Disease
Brief Title: A Study of Recombinant Von Willebrand Factor (rVWF) With or Without ADVATE in Children With Severe Von Willebrand Disease (VWD)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 071102; 2016-001477-33 (EudraCT Number); 2023-509769-18-00 (EU CTIS Number: EU CTR Number)
Record Dates: First submitted 2016-10-12; First posted 2016-10-13 (Estimated); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Von Willebrand Disease
MeSH Terms: conditions — von Willebrand Diseases | interventions — Factor VIII; F8 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- On-demand Treatment (Experimental): Participants will receive vonicog alfa (recombinant von Willebrand factor [rVWF]) treatment for non-surgical bleeding episodes over a 12 to 18-month period.
  Interventions: Biological: Vonicog alfa; Biological: Antihemophilic Factor (Recombinant)
- Elective Surgery (Experimental): 12-24 hours prior to surgery and within 3 hours of surgery. Minor surgery: infuse every 12-24 hours for at least 48 hours based on post-operative dosing. Oral Surgery: infuse at least once within first 8-12 hours post-surgery based on post-operative dosing. Major Surgery: infuse every 12-24 hours for at least first 96 hours post-surgery based on post-operative dosing.
  Interventions: Biological: Vonicog alfa; Biological: Antihemophilic Factor (Recombinant)
- Emergency Surgery (Experimental): Within 3 hours prior to surgery. Minor surgery: infuse every 12-24 hours for at least 48 hours based on post-operative dosing. Oral Surgery: infuse at least once within first 8-12 hours post-surgery based on post-operative dosing. Major Surgery: infuse every 12-24 hours for at least first 96 hours post-surgery based on post-operative dosing.
  Interventions: Biological: Vonicog alfa; Biological: Antihemophilic Factor (Recombinant)

INTERVENTIONS:
Biological: Vonicog alfa — Lyophilized powder and solvent to prepare solution for injection.
  Other Names: VONVENDI; rVWF; BAX 111; TAK-577; SHP677
Biological: Antihemophilic Factor (Recombinant) — Packaged in single boxes with 2 glass vials, with one vial containing the lyophilized ADVATE and the second vial containing the diluent.
  Other Names: Recombinant Factor VIII; rFVIII; Octocog alfa

SUMMARY:
The main aim of the study is to check effectiveness, side effects, and tolerability of vonicog alfa (recombinant von Willebrand factor [rVWF]), with or without ADVATE, in the treatment and control of nonsurgical bleeding events in pediatric participants (less than (<)18 years of age) with severe hereditary von Willebrand disease (VWD).

The participants will be treated with vonicog alfa for 12-18 months. Their von Willebrand Disease will be treated by their doctor according to their doctor's usual clinical practice. During the study, participants will be followed up at clinics or over telephone calls.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of severe von Willebrand disease (VWD) (defined as von Willebrand factor: ristocetin cofactor [VWF:RCo] less than [<] 20 percent [%]):

  * Type 1 (VWF:RCo <20 International Units per deciliter [IU/dL]); or
  * Type 2A (VWF:RCo <20 IU/dL), Type 2B (as diagnosed by genotype), Type 2N (Factor VIII coagulation activity [FVIII:C] <10 % and historically documented genetics), Type 2M; or
  * Type 3 (VWF:Ag less than or equal to [=<] 3 IU/dL).
* Age 0 to <18 years at the time of Screening.
* The participant has provided assent (if appropriate) and legally authorized representative(s) has provided informed consent.
* If female of childbearing potential, participant presents with a negative serum pregnancy test.
* If applicable, participant agrees to employ adequate birth control measures for the duration of the study.
* The participant and/or the legally authorized representative are willing and able to comply with the requirements of the protocol, which should also be confirmed based on a pre-screening evaluation held between the Investigator and the Sponsor, to ensure no eminent risk is present that could challenge the participants compliance with the study requirements.

Additional inclusion criteria for both previously treated participants and participants undergoing surgery are as follows:

* Unable to tolerate are inadequately responsive to, or not a good candidate for 1-deamino-8-D-arginine vasopressin (DDAVP). Examples of participants who are not good candidates for DDAVP include participants with type 2B or type 3 VWD.
* The participant has had a minimum of 1 documented bleed requiring VWF coagulation factor replacement therapy (i.e. treatment with a VWF product) during the previous 12 months prior to enrollment and overall historically 3 or more exposure days (EDs) to VWF replacement therapy.

Additional inclusion criterion for previously untreated participants are as follows:

- The participant has not received prior VWF coagulation factor replacement therapy.

Exclusion Criteria:

* Diagnosis of pseudo-VWD or another hereditary or acquired coagulation disorder (eg, qualitative and quantitative platelet disorders or elevated prothrombin time [PT]/international normalized ratio [INR] greater than [>] 1.4).
* History or presence of a VWF inhibitor at Screening.
* History or presence of a Factor VIII (FVIII) inhibitor with a titer greater than or equal [>=] 0.4 Bethesda units (BU) (by Nijmegen assay) or >=0.6 BU (by Bethesda assay).
* Documented history of a VWF: RCo half-life <6 hours.
* Known hypersensitivity to any of the components of the study drug, such as mouse or hamster proteins.
* Medical history of immunological disorders, excluding seasonal allergic rhinitis/conjunctivitis/asthma, food allergies, or animal allergies.
* Medical history of a thromboembolic event.
* Human immunodeficiency virus (HIV) positive, with an absolute CD4 count <200/ cubic millimeter (mm^3).
* In the judgment of the Investigator, the participant has another clinically significant concomitant disease (e.g. uncontrolled hypertension, cancer) that may pose additional risks for the participant.
* Diagnosis of significant liver disease, as evidenced by, but not limited to, any of the following: serum alanine aminotransferase (ALT) of 5 times the upper limit of normal; hypoalbuminemia; portal vein hypertension (e.g. presence of otherwise unexplained splenomegaly, history of esophageal varices) or liver cirrhosis classified as Child B or C.
* Diagnosis of renal disease, with a serum creatinine level >=2.5 milligram per deciliter (mg/dL).
* Immunomodulatory drug treatment other than anti-retroviral chemotherapy (e.g. α-interferon, or corticosteroid agents at a dose equivalent to hydrocortisone greater than 10 milligram per day [mg/day] (excluding topical treatment [e.g. ointments, nasal sprays]), within 30 days prior to signing the informed consent (or assent, if appropriate).
* If female, participant is pregnant or lactating at the time informed consent (or assent, if appropriate) is obtained.
* Participant has participated in another clinical study involving an investigational product (IP), other than vonicog alfa with or without ADVATE, or investigational device within 30 days prior to enrollment or is scheduled to participate in another clinical study involving an IP other than vonicog alfa or investigational device during the course of this study.
* Participant's legal representative is a family member or employee of the Investigator.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Estimated)
Dates: Start 2017-11-06 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Hemostatic Efficacy | Within 24 hours after the last infusion of study drug following the onset of the bleeding episode (if/when the severity and/or duration of the bleeding requires the infusion of the study drug)
  Treatment success for vonicog alfa-treated nonsurgical bleeding episodes (using a 4-point scale: Excellent, Good, Moderate, None).

SECONDARY OUTCOMES:
Number of Treated Nonsurgical Bleeding Episodes With an Efficacy Rating of 'Excellent' or 'Good' | Throughout the study duration of approximately 8.5 years
  If/when the severity and/or duration of the bleeding requires the infusion of the study drug.
Number of Infusions per Bleeding Episode | Throughout the study duration of approximately 8.5 years
Number of Vonicog Alfa Units per Bleeding Episode | Throughout the study duration of approximately 8.5 years
Number of ADVATE Units (if needed) per Bleeding Episode | Throughout the study duration of approximately 8.5 years
Elective or Emergency Surgery: Assessment of Hemostatic Efficacy - Immediately After Surgery | Immediately after surgery
  Assessed by the operating surgeon, based on a 4-point ordinal scale: Excellent, Good, Moderate, None.
Elective or Emergency Surgery: Overall Assessment of Hemostatic Efficacy 24 Hours After the Last Perioperative Infusion of rVWF | 24 hours after last perioperative rVWF infusion
  Assessed by the Investigator (hematologist) on a 4-point ordinal scale: Excellent, Good, Moderate, None.
Elective or Emergency surgery: Overall Assessment of Hemostatic Efficacy Day 7 Post-operative | Post-operative Day 7
  Assessed by the Investigator (hematologist) on a 4-point ordinal scale: Excellent, Good, Moderate, None.
Elective or Emergency surgery: Overall Assessment of Hemostatic Efficacy Day 14 Post-operative | Post-operative Day 14
  Assessed by the Investigator (hematologist) on a 4-point ordinal scale: Excellent, Good, Moderate, None.
Incidence and Severity of Adverse Events (AEs) | Throughout the study period of approximately 8.5 years
Incidence of Thromboembolic Events | Throughout the study period of approximately 8.5 years
Incidence of Severe Hypersensitivity Reactions | Throughout the study period of approximately 8.5 years
Development of Neutralizing Antibodies to von Willebrand Factor (VWF) and Factor VIII (FVIII) | Throughout the study period of approximately 8.5 years
Development of Total Binding Antibodies to von Willebrand Factor (VWF) | Throughout the study period of approximately 8.5 years
Development of Antibodies to Chinese Hamster Ovary (CHO) Proteins, Murine Immunoglobulin G (IgG), and rFurin | Throughout the study period of approximately 8.5 years
Area Under the Plasma Concentration/Time Curve From 0 to 96 Hours Post-Infusion (AUC0-96h) for Von Willebrand factor: ristocetin cofactor (VWF:Rco), von Willebrand factor: antigen (VWF:Ag) and von Willebrand factor: collagen binding capacity (VWF:CB) | Within 30 minutes prior to infusion and post infusion at: SEQUENCE 1: 1, 24, 72 hours; SEQUENCE 2: 0.25, 12, and 48 hours; SEQUENCE 3: 6, 30, and 96 hours
Area Under the Plasma Concentration/Time Curve From Time 0 to Infinity (AUC0-inf) for VWF:RCo, VWF:Ag and VWF:CB | Within 30 minutes prior to infusion and post infusion at: SEQUENCE 1: 1, 24, 72 hours; SEQUENCE 2: 0.25, 12, and 48 hours; SEQUENCE 3: 6, 30, and 96 hours
Mean Residence Time (MRT) for VWF:RCo, VWF:Ag and VWF:CB | Within 30 minutes prior to infusion and post infusion at: SEQUENCE 1: 1, 24, 72 hours; SEQUENCE 2: 0.25, 12, and 48 hours; SEQUENCE 3: 6, 30, and 96 hours
Time to Reach Maximal Plasma Concentration (Tmax) for VWF:RCo, VWF:Ag and VWF:CB | Within 30 minutes prior to infusion and post infusion at: SEQUENCE 1: 1, 24, 72 hours; SEQUENCE 2: 0.25, 12, and 48 hours; SEQUENCE 3: 6, 30, and 96 hours
Maximal Plasma Concentration (Cmax) for VWF:RCo, VWF:Ag and VWF:CB | Within 30 minutes prior to infusion and post infusion at: SEQUENCE 1: 1, 24, 72 hours; SEQUENCE 2: 0.25, 12, and 48 hours; SEQUENCE 3: 6, 30, and 96 hours
Clearance (CL) for VWF:RCo, VWF:Ag and VWF:CB | Within 30 minutes prior to infusion and post infusion at: SEQUENCE 1: 1, 24, 72 hours; SEQUENCE 2: 0.25, 12, and 48 hours; SEQUENCE 3: 6, 30, and 96 hours
Incremental Recovery (IR) for VWF:RCo, VWF:Ag and VWF:CB | Within 30 minutes prior to infusion and post infusion at: SEQUENCE 1: 1, 24, 72 hours; SEQUENCE 2: 0.25, 12, and 48 hours; SEQUENCE 3: 6, 30, and 96 hours
In-vivo Recovery (IVR) for VWF:RCo, VWF:Ag and VWF:CB | Within 30 minutes prior to infusion and post infusion at: SEQUENCE 1: 1, 24, 72 hours; SEQUENCE 2: 0.25, 12, and 48 hours; SEQUENCE 3: 6, 30, and 96 hours
Elimination Phase Half-life (T1/2) for VWF:RCo, VWF:Ag and VWF:CB | Within 30 minutes prior to infusion and post infusion at: SEQUENCE 1: 1, 24, 72 hours; SEQUENCE 2: 0.25, 12, and 48 hours; SEQUENCE 3: 6, 30, and 96 hours
Volume of Distribution at Steady State (Vss) for VWF:RCo, VWF:Ag and VWF:CB | Within 30 minutes prior to infusion and post infusion at: SEQUENCE 1: 1, 24, 72 hours; SEQUENCE 2: 0.25, 12, and 48 hours; SEQUENCE 3: 6, 30, and 96 hours
Area Under the Plasma Concentration/Time Curve From 0 to 96 Hours Post-infusion (AUC0-96h) for Factor VIII (FVIII) Activity | Within 30 minutes prior to infusion and post infusion at: SEQUENCE 1: 1, 24, 72 hours; SEQUENCE 2: 0.25, 12, and 48 hours; SEQUENCE 3: 6, 30, and 96 hours

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (46):
- United States (16):
  - University of Colorado Hemophilia & Thrombosis Center, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida College of Medicine, Jacksonville, Florida
  - Bleeding and Clotting Disorders Institute, Peoria, Illinois
  - Indiana Hemophilia and Thrombosis Center, Indianapolis, Indiana
  - University of Nebraska Medical Center, Omaha, Nebraska
  - St. Jude Affiliate Clinic at Novant Health, Charlotte, North Carolina
  - Comprehensive Cancer Center of Wake Forest Unversity, Winston-Salem, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Texas Children's Cancer and Hematology Center, Houston, Texas
  - Texas Children's Hospital, Houston, Texas
  - Comprehensive Center for Bleeding Disorders, Milwaukee, Wisconsin
- Austria (2):
  - Medizinische Universität Innsbruck, Innsbruck
  - AKH - Medizinische Universität Wien, Vienna
- UZ Leuven, Leuven, Belgium
- Fakultni nemocnice Brno, Brno, Czechia
- France (8):
  - Hôpital Morvan, Brest, Finistere
  - Groupe Hospitalier Pellegrin - Hôpital Pellegrin, Bordeaux
  - Groupement Hospitalier Est- Hôpital Louis Pradel, Bron
  - CHU CAEN - Hôpital de la Côte de Nacre, Caen
  - Groupement Hospitalier Sud - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Hopital Cardiologique - CHU Lille, Lille
  - CHU de Nantes Site Hotel Dieu, Nantes
  - Hôpital Necker - Enfants Malades, Paris
- Germany (3):
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Werlhof-Institut GmbH, Hanover
  - Medizinische Hochschule Hannover, Hanover
- Italy (4):
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Fondazione IRCCS CA' Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliera Pediatrica Santobono Pausillipon, Napoli
  - Ospedale Pediatrico Bambino Gesù, Roma
- Erasmus Medisch Centrum, Rotterdam, Netherlands
- Russia (3):
  - SBEI HPE Altai State Medical University of MoH and SD, Barnaul
  - SAIH "Kemerovo Regional Clinical Hospital", Kemerovo
  - FSBI of Science "Kirov Scientific and Research Institute of Hematology and Blood Transfusion of FMBA, Kirov
- Spain (2):
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitari i Politecnic La Fe, Valencia
- Turkey (Türkiye) (3):
  - Istanbul University Cerrahpasa Medical Faculty, Istanbul
  - Ege University Medical Faculty, Izmir
  - Ondokuz Mayis Univ. Med. Fac., Samsun
- SI Institute of Blood Pathology and Transfusion Medicine of NAMSU, Lviv, Ukraine
- Royal Manchester Children's Hospital, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fc34db2bf003ab45926